CLINICAL TRIAL: NCT03776279
Title: Single-arm, Open and Multi-center Phase II Study of Liposome-entrapped Mitoxantrone Hydrochloride Injection in Relapsed/Refractory Peripheral T-cell Lymphoma and NK/T-cell Lymphoma
Brief Title: A Study of Liposome-entrapped Mitoxantrone Hydrochloride Injection in Relapsed/Refractory Peripheral T-cell Lymphoma and NK/T-cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLM60-PTCL
Record Dates: First submitted 2018-12-13; First posted 2018-12-14 (Actual); Last update posted 2018-12-14 (Actual); Status verified 2018-12

CONDITIONS: Relapsed or Refractory Peripheral T-cell and NK/T-cell Lymphoma
MeSH Terms: conditions — Recurrence; Lymphoma, Extranodal NK-T-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mitoxantrone Hydrochloride Liposome Injection (Experimental): 4 weeks is a treatment cycle, and the first day of each cycle is administered.
  Interventions: Drug: Mitoxantrone Hydrochloride Liposome Injection

INTERVENTIONS:
Drug: Mitoxantrone Hydrochloride Liposome Injection — Mitoxantrone Hydrochloride Liposome Injection 20 mg/m2 will be infused intravenously once over 60min in 250 ml 5％ glucose injection on the first day during a treatment phase of 4 weeks.

SUMMARY:
This is a single-arm, open, multi-center, phase II study to evaluate the efficacy and safety of Mitoxantrone Hydrochloride Liposome Injection in Relapsed or refractory peripheral t-cell and NK/T-cell lymphoma.

DETAILED DESCRIPTION:
The dosage regimen of Liposome-entrapped Mitoxantrone is multi-cycle 20mg/m2 intravenous infusion. Every 4 weeks is a treatment cycle, with administration on the first day of each cycle. End-of-treatment visit will be made to the subjects within 4 weeks after the end of the last administration. Progression-free survival (PFS) follow-up will be conducted to the subjects in stable or improved condition after treatment and the subjects with early termination of treatment due to intolerance in Week 8 after the last administration of study drug, and thereafter once every 8 weeks until PD, death, withdrawal of informed consent form (ICF), starting another new treatment or end of the entire study (whichever occurs first). Meanwhile, overall survival (OS) follow-up will also be conducted to the subjects with PD and starting another new treatment once every 8 weeks until death, withdrawal of ICF or end of the entire study (whichever occurs first).

ELIGIBILITY:
Inclusion criteria

Subjects must satisfy all the following conditions before enrollment:

1. Those who have fully understood the study and have signed the ICF.
2. Male or female, aged 18 or above (including 18).
3. Those with PTCL and NK/T-cell lymphoma confirmed by histopathological and/or cytological examination, with the subtypes as follows:

   1. Peripheral T-cell lymphoma, unspecified (PTCL, NOS)
   2. Angioimmunoblastic T-cell lymphoma (AITL)
   3. ALK+systematic anaplastic large T-cell lymphoma (ALCL, ALK+)
   4. ALK-systematic anaplastic large T-cell lymphoma (ALCL，ALK-)
   5. Extranobal NK/T cell lymphoma (nasal type) (NKTCL)
   6. Enteropathy-associated T-cell lymphoma (EATCL, Type I (traditional type), Type II)
   7. Hepatosplenic γδ T-cell lymphoma (HSTCL, γδT) hOther non-Hodgkin's lymphomas from invasive T-cells (other than highly invasive cells) approved by the sponsor, who may be enrolled in the opinion of the investigator.
4. Those receivd at least first-line standard treatment (including chemotherapy and autologous hematopoietic stem cell transplantation) If anthracycline or anthracycline-containing chemotherapy has been used in the past, the efficacy is assessed as response; if they were NK/T-cell lymphoma patients, they need to be treated with asparaginase (or pepsinase, L-asparaginase) treatment.
5. Subjects who must provide the written pathological/histological diagnosis report during the screening period, and agree to provide the tumor tissue sections or fresh tumor tissues to the Center Laboratory for testing.
6. Those with ECOG performance status score of 0 or 1.
7. The estimated survival time was at least 12 weeks.
8. Those at least with one measurable lesion in accordance with the revised standard for evaluation of efficacy in malignant lymphoma (Version 2007): the long axis of the lesion shall be>1.5 cm or 1.0~1.5 cm and the short axis of the lesion shall be>1.0 cm.
9. Subjects who shall meet the following requirements for laboratory examination when screening and who have not received cell growth factor (long-acting granulocyte-colony stimulating factor [G-CSF] and [PEG-CSF] shall have the interval of 14 days) and platelet or granulocyte infusion within 7 days before hematological evaluation for screening:

   1. Absolute value of neutrophils ≥ 1.5 × 109/ L in subjects without involvement of bone marrow; absolute value of neutrophil ≥ 1.0 × 109/ L in subjects with involvement of bone marrow;
   2. Hemoglobin ≥ 90 g/L (without red cell infusion within 14 days), hemoglobin ≥ 75 g/ L in subjects with involvement of bone marrow;
   3. Platelet ≥ 75 × 109/ L in subjects without involvement of bone marrow; platelet ≥ 50 × 109/ L in subjects with involvement of bone marrow;
   4. Serum total bilirubin ≤ 1.5 × upper limit of normal (ULN) (total bilirubin ≤ 3 × ULN if bilirubin level increase is caused by lymphoma invading the liver);
   5. Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 2.5 × ULN; if AST or ALT increase is caused by lymphoma invading the liver, both AST and ALT shall be ≤ 5 × ULN);
   6. Creatinine < 1.5 × ULN.
10. Female subjects:

    1. Without fertility (i.e., unable to get pregnant under physiological condition), including postmenopausal (complete cessation of menstruation for ≥ 1 year) or documented irreversible sterilization including hysterectomy, bilateral ovariectomy or bilateral salpingectomy (rather than tubal ligation);
    2. With fertility potential, who shall be negative when serum pregnancy test screening (within 7 days of the first administration of study drug) and agree to take effective contraception measures during the study period and within 90 days after the last administration. Subjects shall always practice contraception strictly in accordance with the labels of contraceptive drugs/devices and the instructions of the investigator. Effective contraception measures shall be defined as follows:

    i)Sex partner vasectomized is the sole sex partner of the female subject; ii)Use of IUDs with a failure rate of less than 1% per year iii)Double contraception, e.g. spermatocide plus male condom, female condom, diaphragm, cervical cap or intrauterine device.

    Male subjects: who shall have received the vasectomy, or agree to take effective contraception measures during the study period and within 30 days after the last administration.
11. Subjects who are able to comply with the study procedures, restrictions and requirements as judged by the investigator.

Exclusion criteria

Subjects consistent with any one of the following conditions:

1. Subjects in lymphoma leukemia (malignant cell proportion of > 20% in bone marrow examination);
2. Subjects are consistent with one of the following conditions in the previous anti-tumor treatment history:

   1. Those receiving Mitoxantrone or Liposome-entrapped Mitoxantrone previously;
   2. Those receiving treatment of Adriamycin or other anthracyclines previously, with the total cumulative dose of > 360 mg/m2 (when converted to 1 mg Adriamycin, other anthracyclines shall be equivalent to 2 mg Epirubicin or 2 mg Pirarubicin or 2 mg Daunorubicin or 0.5 mg Idarubicin);
   3. Those receiving anti-tumor treatment (including chemotherapy, radiotherapy, hormone therapy or administration of TCM with anti-tumor activity) within 4 weeks prior to the first use of the study drug);
   4. Those receiving autologous hematopoietic stem cell transplantation within 6 months;
   5. Those receiving allogeneic hematopoietic stem cell transplantation previously.
3. Those receiving major surgery (the definition of major surgery shall refer to the Level 3 or 4 surgery stipulated in the Management Practices of Clinical Application of Medical Technology) within 4 weeks prior to enrollment or those who have not completely recovered from any previous invasive operation.
4. Those who have not recovered from toxic response in the previous anti-tumor treatment (>Grade 1 in NCI-CTCAE [Version 4.03], with the exception of hair loss and pigmentation.
5. Those with other malignant tumors previously or currently (except the non-melanoma skin basal cell carcinoma under effective control, breast/cervical carcinoma in situ, and other malignant tumors not treated but under effective control in the past five years).
6. Subjects with known or existing primary or metastatic central nervous system lymphoma, or with existing other cerebral/meningeal diseases.
7. Subjects with uncontrolled hypertension (refers to systolic pressure of 180 mmHg and/or diastolic pressure of 100 mmHg after treatment).
8. Subjects with active hemorrhagic disease.
9. Subjects with active infection, including hepatitis B (positive hepatitis B virus surface antigen and hepatitis B virus DNA of more than 1,000 copies/mL) and hepatitis C (positive hepatitis C virus RNA).
10. Human immunodeficiency virus (HIV) infection (HIV positive).
11. Subjects with history of hepatic fibrosis or cirrhosis or with clinical signs and symptoms suggestive of liver fibrosis or cirrhosis.
12. Subjects with the cardiac function and disease:

    1. Male: QTc>450 ms, female: QTc>470 ms when ECG examination in the Research Center during the screening period;
    2. Clinically significant arrhythmias, including but not limited to complete left bundle branch block, Degree II atrioventricular block and PR interval > 250 ms;
    3. Any risk factor that might increase the QTc interval, e.g. hypokalaemia, inherited long-QT syndrome, with current administration of the drug for prolonging the QT interval or discontinuance for less than 15 days;
    4. Congestive heart failure of ≥Grade 2 in the New York Heart Association;
    5. Cardiac ejection fraction less than 50% or less than the lower limit of laboratory examination vale range of Research Center;
    6. Within six months prior to recruitment occurred myocardial infarction, unstable angina, severe unstable ventricular arrhythmia or any other arrhythmia requiring treatment, clinical history of severe pericardial disease, or electrocardiographic evidence of acute ischemia or abnormal active conduction system.
13. Subjects with known history of immediate or delayed hypersensitivity to the similar drug and excipient of the study drug.
14. Pregnant or lactating women.
15. According to the judgement of the investigators ,Those with any severe or uncontrolled systematic disease, systematic complication, other severe complicated diseases (e.g. hemophagocytic syndrome) or special tumor condition that might make the subjects unsuitable for entry into the study or might affect the compliance to the protocol or might cause significant interference with the correct evaluation of safety, toxicity and efficacy of the study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2018-04-02 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | >4weeks
  The percentage of complete response (CR) and partial response (PR) in all the enrolled subjects from the date of the first administration (calculated by the optimum response during the entire study period)

SECONDARY OUTCOMES:
Duration of Response(DoR) | >3 months
  The duration from achieving effective treatment (CR or PR recorded for the first time) until definite relapse or progression for the first time.
Progression-free survival(PFS) | 3 years
  The duration from the first administration date until lymphoma progression (PD evaluated by imaging diagnosis) date or all-cause death date (whichever occurs first).
Overall survival(OS) | 3 years
  The duration from the first administration date until all-cause death date.
Disease control rate(DCR) | 3 years
  The percentage of CR and PR in all the enrolled subjects from the date of the first administration, including the subjects with CR, PRC or SD

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China